CLINICAL TRIAL: NCT04954716
Title: Comparison of Deep Friction Massage and Post Isometric Relaxation Technique in Cervicogenic Headache
Brief Title: Manual Techniques in Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/20/0111/Bushra
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic headache (CH, CGH); Muscle Energy Technique (MET); ,Post-isometric relaxation(PIR)
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep Neck Flexor Massage (Experimental): INTERVENTIONAL GROUP(DEEP Neck FLEXOR MASSAGE)
  Interventions: Other: Deep Neck Flexor Massage
- Post-Isometric Relaxation Technique (Active Comparator): CONTROL GROUP (POST-ISOMETRIC RELAXATION TECHNIQUE)
  Interventions: Other: Post-Isometric Relaxation Technique

INTERVENTIONS:
Other: Deep Neck Flexor Massage — Deep friction massage is a specific connective tissue massage that was given across the affected fibers.The therapist's fingers and patient's skin must move as one, otherwise moving subcutaneous fascia against muscle or ligament could lead to blister formation or subcutaneous bruising.The friction massage must have sufficient sweep and be deep enough.
  Arms: Deep Neck Flexor Massage
Other: Post-Isometric Relaxation Technique — The PIR technique is performed as follows.The hypertonic muscle is taken to a length just short of pain, or to the point where resistance to movement is first noted.A submaximal (10-20%) contraction of the hypertonic muscle is performed away from the barrier for between 5 and 10 seconds and the therapist applies resistance in the opposite direction . The patient should inhale during this effort.After the isometric contraction the patient is asked to relax and exhale while doing so.Following this a gentle stretch is applied to take up the slack till the new barrier.Starting from this new barrier, the procedure is repeated two or three times.
  Arms: Post-Isometric Relaxation Technique

SUMMARY:
This project will explore the effect of deep friction massage and post isometric relaxation techniques in Cervicogenic headache. The population sample will be 20 divided randomly into two groups by Lottery method. Then i will collect data from central hospital, Gujranwala. One group will be treated with a deep friction massage technique thrice a week for 3 weeks. Another group will be treated with a post isometric relaxation technique thrice a week for 3 weeks. Both groups will receive a heating pad and neck isometric as baseline treatment. Baseline measurements are taken by an inclinometer. After a treatment plan, the group will be assessed again and post-treatment measured values will be compared with the pretest values. Subjects will be asked to come for follow-up after 4 weeks. The follow-up will show which technique is more effective in subjects having Cervicogenic headaches. Both the techniques used are non-invasive and having minimum side effects. This project will help Physical Therapy Practitioner to explore which technique is more useful to treat Cervicogenic headaches.

DETAILED DESCRIPTION:
Cervicogenic headache is a relatively common and still controversial form of headache arising from structures in the neck. In patients with this disorder, attacks or chronic fluctuating periods of neck/head pain may be provoked by the sustained neck. The International Headache Society (IHS), 2013 defined Cervicogenic Headache (CGH) as a secondary headache, which implies that headache is caused by a disorder of the cervical spine and its components bony, disc, and soft tissue elements. CGH can be a perplexing pain disorder that is refractory to treatment if it is perceived. Patients with CGH exhibited decreases in the quality of life comparable to migraine patients and patients with tension-type headaches, with even lower scores for physical functioning.

.Headache is a common disorder affecting up to 66% of the general population. headache negatively influences both quality of life and labor productivity.Cervicogenic headache is one of the common types of headache accounting for 0.4-15% of the headache population.

we distinguished it from other types of headaches, such as a migraine, that may present with some common symptoms. The International Headache Society (IHS) classified CGH as a secondary headache arising from musculoskeletal disorders in the cervical spine. The complicated convergence of cervical afferents with trigeminal afferents in the trigemino-cervical complex is intended as the physiologic basis of a headache arising from cervical structures.

The aim of friction massage is to take care of the quality at intervals the soft tissue structures of ligament, tendon, and muscle and stop adherent scars from forming. The massage is deep and should be applied transversally to the precise tissue concerned in contrast to the superficial massage given within the longitudinal direction parallel to the vessels which boosts circulation and come of fluid. Profound cervical flexor (DCF) has a noteworthy postural capacity in supporting and rectifying the cervical lordosis. It has been discovered that specific muscles in the cervical spine have a tendency to debilitate , the most widely recognized of these being the DCF.

MET is a treatment technique that includes a willful constriction of a subject's muscle in a correctly controlled bearing, against a counterforce that is given by the specialist. MET is utilized to diminish the pain, extend the tight muscles and belts, decrease muscle tone, enhances nearby flow, strengthen the feeble musculature, and mobilizes the joint restrictions. MET increases the extensibility of muscles and spinal range of motion, treating patients with reduced mobility. Extending includes the use of manual or mechanical power to prolong/protract the structures that are adaptively been abbreviated and are hypomobile.

Post-isometric relaxation (PIR) may be a technique typically employed by manual therapists for treating muscle tension and joint pathology in myofascial pain syndromes There is a lack of evidence demonstrating the efficacy of deep friction massage therapy in the management of cervicogenic headache, particularly targeting cervical muscle tightness related to Cervicogenic headache. The purpose of this study is to compare the effect of soft tissue massage with MET to access which technique has a greater clinical impact than others in improving cervicogenic headache.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Symptoms duration more than 6 months.
* Age 18 -60
* Patient has confirmed the diagnosis of cervicogenic headache

Exclusion Criteria:

* Rule out cervical malignancy
* infection (such as osteomyelitis or diskitis)
* osteoporosis, inflammatory arthritis.
* fracture, pregnancy
* cord compression, uncontrolled hypertension
* cardiovascular disease
* in the setting of carotid or vertebral artery disease.
* Trauma cases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Headache disability index | 3 week
  This scale is used to identify difficulties that you may be experiencing because of your headache. Please check off "YES", "SOMETIMES", or "NO" to each item. Proforma consist of 25 question
  Scoring The following responses are given the following values:
  Response Points Yes 4 Sometimes 2 No 0 Interpretation A 29 point change (95% confidence interval) or greater in the total score from test to retest must occur before the change can be attributed to treatment effects.

SECONDARY OUTCOMES:
Upper cervical spine(ROM) | 3 weeks
  standard technique for measuring cervical spine motions in different rotations, including sagittal, frontal, transversal, and rotational

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sana ullah, MS, Principal Investigator — Riphah International University
Locations (1):
- Central hospital Gujranwala, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martelletti P, van Suijlekom H. Cervicogenic headache: practical approaches to therapy. CNS Drugs. 2004;18(12):793-805. doi: 10.2165/00023210-200418120-00004. PMID 15377169
- [Background] Stovner Lj, Hagen K, Jensen R, Katsarava Z, Lipton R, Scher A, Steiner T, Zwart JA. The global burden of headache: a documentation of headache prevalence and disability worldwide. Cephalalgia. 2007 Mar;27(3):193-210. doi: 10.1111/j.1468-2982.2007.01288.x. PMID 17381554
- [Background] Castien RF, De Hertogh W, Scholten-Peeters GG. Letter to the Editor: Physical examination tests for screening and diagnosis of cervicogenic headache: A systematic review by Rubio-Ochoa et al. (2015). Man Ther. 2016 Jun;23:e7-8. doi: 10.1016/j.math.2016.01.006. Epub 2016 Jan 29. No abstract available. PMID 26934859
- [Background] Fernandez-de-Las-Penas C, Alonso-Blanco C, Cuadrado ML, Pareja JA. Spinal manipulative therapy in the management of cervicogenic headache. Headache. 2005 Oct;45(9):1260-3. doi: 10.1111/j.1526-4610.2005.00253_1.x. PMID 16178960
- [Background] Garcia JD, Arnold S, Tetley K, Voight K, Frank RA. Mobilization and Manipulation of the Cervical Spine in Patients with Cervicogenic Headache: Any Scientific Evidence? Front Neurol. 2016 Mar 21;7:40. doi: 10.3389/fneur.2016.00040. eCollection 2016. PMID 27047446
- [Background] Bogduk N. Cervicogenic headache: anatomic basis and pathophysiologic mechanisms. Curr Pain Headache Rep. 2001 Aug;5(4):382-6. doi: 10.1007/s11916-001-0029-7. PMID 11403743
- [Background] Li L, Stoop R, Clijsen R, Hohenauer E, Fernandez-de-Las-Penas C, Huang Q, Barbero M. Criteria Used for the Diagnosis of Myofascial Trigger Points in Clinical Trials on Physical Therapy: Updated Systematic Review. Clin J Pain. 2020 Dec;36(12):955-967. doi: 10.1097/AJP.0000000000000875. PMID 32841969
- [Background] Chamberlain GJ. Cyriax's Friction Massage: A Review. J Orthop Sports Phys Ther. 1982;4(1):16-22. doi: 10.2519/jospt.1982.4.1.16. PMID 18810110
- [Background] Emary P. Use of post-isometric relaxation in the chiropractic management of a 55-year-old man with cervical radiculopathy. J Can Chiropr Assoc. 2012 Mar;56(1):9-17. PMID 22457537
- [Background] Youssef EF, Shanb AS. Mobilization versus massage therapy in the treatment of cervicogenic headache: a clinical study. J Back Musculoskelet Rehabil. 2013;26(1):17-24. doi: 10.3233/BMR-2012-0344. PMID 23411644
- [Background] Chaibi A, Russell MB. Manual therapies for cervicogenic headache: a systematic review. J Headache Pain. 2012 Jul;13(5):351-9. doi: 10.1007/s10194-012-0436-7. Epub 2012 Mar 30. PMID 22460941